CLINICAL TRIAL: NCT01686139
Title: Phase 1 Study: Treatment of Patients With Diabetic Foot Complications With Allogeneic Bone Marrow Derived Mesenchymal Stromal Cells (ABMD-MSC)
Brief Title: Safety Study of Stem Cells Treatment in Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Itzhak Siev-Ner, Head of the Orthopedic Rehabilitation Department, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-11-8802-IS-SMC
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Type I Diabetes Mellitus With Ulcer; Type II Diabetes Mellitus With Ulcer
Keywords: Diabetic mellitus; Diabetic foot ulcers; Ischemic Limb
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABDM-MSC (Experimental): The patient will receive multiple injections in one session during the study. The injections will take place in the chronic wound bed and in the third distal part of the treated shin (in the form of a ring).
  Maximal amount of ABMD-MSC cells injected: 10-20*10^6 cells (up to volume of 20mL, depending on the wound size & patient weight).
  Interventions: Biological: ABMD-MSC

INTERVENTIONS:
Biological: ABMD-MSC — 10-20 x 10^6 cells/20mL

SUMMARY:
Diabetes Mellitus (DM) can be regarded as one of the "epidemics" of the western world.

DM contributes to severe morbidity and mortality due to damage in the target organs (neuropathy, vasculopathy, nephropathy, retinopathy).

It affects the quality of life of the patients because of increased rate of blindness, IHD, stroke, end stage renal failure, hemodialysis and lower limb amputations (LLA).The Diabetic Foot (DF) is defined as destruction or infection of tissue/s in the foot of diabetic patients due to neurological damage and / or different levels of Peripheral Vascular Disease (PVD). Diabetic foot complications are the most common cause of lower extremity amputations in the industrialized world. The lifetime occurence of Diabetic Foot Ulcers (DFU) is 20% in diabetic patients.

Between 15% - 25% of the foot ulcers will lead to lower limb amputations.

It has been shown that Mesenchymal Stem Cells (MSCs) could be an effective therapy for many diseases including acute respiratory distress syndrome, spinal cord injury, liver injury and critical limb ischemia.

Stem cells can be obtained from either the patient (autologous) or non-related healthy donors (allogeneic).

The purpose of this study is to determine the safety and efficacy of cultured Bone Marrow Mesenchymal Stromal Cells (BM-MSCs) from allogeneic donors for treatment of chronic leg wounds of diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient signed informed consent.
* Adult males or females between 18 and 81 years of age with diabetes mellitus type 1 or type 2.
* Patient has one Diabetic Foot Ulcer (DFU) on the treated leg. The size of the DFU is no greater than 10 cm2 .
* The Diabetic Foot Ulcer (DFU) is neuropathic: The patient is checked by a 5.27 mm Monofilament, and doesn't have a sensation in at least 4 of 9 points in the foot.
* No endovascular or surgical interventions are planned.
* Patient isn't in an immediate life threat.
* Normal organ and marrow function as defined:

  1. Leukocytes ≥3,000/μL
  2. Absolute neutrophil count ≥1,500/μL
  3. Platelets ≥140,000/μL
  4. AST (SGOT)/ALT (SGPT) ≤2.5 X institutional standards range
  5. Creatinine ≤ 2.5 mg/dL
* Patients with controlled blood pressure (defined as a systolic blood pressure ≤180 and/or a diastolic blood pressure of ≤110 mmHg) and established anti-hypertensive therapy as necessary prior to entry into the study.

Exclusion Criteria:

* Patient weight is greater than 120 Kg.
* Patients with poorly controlled diabetes mellitus (HbA1c > 10%).
* Presence of osteomyelitis (stage B grade 3 and stage D grade 3 on the UT Scale).
* More than one ulcer in the treated foot.
* Patients with a known failed ipsilateral revascularization procedure within 4 weeks prior to enrollment.
* Patients with ABI <= 0.3
* Patients receiving treatment with hematopoietic growth factors.
* (Actively) infected ulcer.
* Infection of the involved extremity(ies) in the intended region of injection. Patient will be included (injected) if there is a safe zone of 10 cm from any soft tissue infection, manifested by fever, purulence and severe cellulitis.
* Active wet gangrenous tissue.
* Patients who require uninterrupted anticoagulation or anti-platelet therapy [i.e. anticoagulation therapy (e.g. Coumadin) that cannot be stopped for 72 hours prior to intramuscular injections.
* Patients with a blood clotting disorder not caused by medication.
* Patients with known cancer undergoing treatment including chemotherapy, radiotherapy or immunotherapy.
* Patients with end stage renal disease requiring dialysis.
* Patients who are pregnant or lactating.
* History of regular alcohol consumption exceeding 2 drinks/day (1 drink = 5 oz [150mL] of wine or 12 oz [360mL] of beer or 1.5 oz [45mL] of hard liquor) within 6 months of screening and/or history of illicit drug use.
* Known allergies to protein products (horse or bovine serum, or porcine trypsin) used in the cell production process.
* Patients receiving experimental medications or participating in another clinical study within 30 days of screening.
* Immune deficient patients.
* Patients with positive blood tests for Hepatitis B or Hepatitis C or HIV or Syphilis at the time of screening.
* Patients treated by Ilomedin (Iloprost).
* Patients having received a new chronic pharmacologic treatment regimen within 4 weeks prior to enrollment.
* Patients undergoing hyperbaric oxygen treatment within 4 weeks of inclusion and/or required throughout the trial.
* Concomitant wound treatments that include growth factors or tissue engineered products.
* In the opinion of the investigator, the patient is unsuitable for cellular therapy.
* Patients receiving systemic or direct target limb injection of antiangiogenic drugs.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events | 6 months after treatment
  Frequency and severity of Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Siev-Ner, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Orthopedic Rehabilitation out-patient clinic, Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Friedenstein AJ, Gorskaja JF, Kulagina NN. Fibroblast precursors in normal and irradiated mouse hematopoietic organs. Exp Hematol. 1976 Sep;4(5):267-74. PMID 976387
- [Background] Meirelles Lda S, Fontes AM, Covas DT, Caplan AI. Mechanisms involved in the therapeutic properties of mesenchymal stem cells. Cytokine Growth Factor Rev. 2009 Oct-Dec;20(5-6):419-27. doi: 10.1016/j.cytogfr.2009.10.002. Epub 2009 Nov 18. PMID 19926330
- [Background] Wu Y, Zhao RC, Tredget EE. Concise review: bone marrow-derived stem/progenitor cells in cutaneous repair and regeneration. Stem Cells. 2010 May;28(5):905-15. doi: 10.1002/stem.420. PMID 20474078
- [Background] Sensebe L, Krampera M, Schrezenmeier H, Bourin P, Giordano R. Mesenchymal stem cells for clinical application. Vox Sang. 2010 Feb;98(2):93-107. doi: 10.1111/j.1423-0410.2009.01227.x. Epub 2009 Aug 3. PMID 19663934
- [Background] Chen L, Tredget EE, Wu PY, Wu Y. Paracrine factors of mesenchymal stem cells recruit macrophages and endothelial lineage cells and enhance wound healing. PLoS One. 2008 Apr 2;3(4):e1886. doi: 10.1371/journal.pone.0001886. PMID 18382669
- [Background] Fu X, Fang L, Li X, Cheng B, Sheng Z. Enhanced wound-healing quality with bone marrow mesenchymal stem cells autografting after skin injury. Wound Repair Regen. 2006 May-Jun;14(3):325-35. doi: 10.1111/j.1743-6109.2006.00128.x. PMID 16808812
- [Background] McFarlin K, Gao X, Liu YB, Dulchavsky DS, Kwon D, Arbab AS, Bansal M, Li Y, Chopp M, Dulchavsky SA, Gautam SC. Bone marrow-derived mesenchymal stromal cells accelerate wound healing in the rat. Wound Repair Regen. 2006 Jul-Aug;14(4):471-8. doi: 10.1111/j.1743-6109.2006.00153.x. PMID 16939576
- [Background] Wu Y, Wang J, Scott PG, Tredget EE. Bone marrow-derived stem cells in wound healing: a review. Wound Repair Regen. 2007 Sep-Oct;15 Suppl 1:S18-26. doi: 10.1111/j.1524-475X.2007.00221.x. PMID 17727462
- [Background] Kwon DS, Gao X, Liu YB, Dulchavsky DS, Danyluk AL, Bansal M, Chopp M, McIntosh K, Arbab AS, Dulchavsky SA, Gautam SC. Treatment with bone marrow-derived stromal cells accelerates wound healing in diabetic rats. Int Wound J. 2008 Jun;5(3):453-63. doi: 10.1111/j.1742-481X.2007.00408.x. PMID 18593394
- [Background] Brem H, Tomic-Canic M. Cellular and molecular basis of wound healing in diabetes. J Clin Invest. 2007 May;117(5):1219-22. doi: 10.1172/JCI32169. PMID 17476353
- [Background] Iwase T, Nagaya N, Fujii T, Itoh T, Murakami S, Matsumoto T, Kangawa K, Kitamura S. Comparison of angiogenic potency between mesenchymal stem cells and mononuclear cells in a rat model of hindlimb ischemia. Cardiovasc Res. 2005 Jun 1;66(3):543-51. doi: 10.1016/j.cardiores.2005.02.006. Epub 2005 Mar 2. PMID 15914119
- [Background] Rafii S, Lyden D. Therapeutic stem and progenitor cell transplantation for organ vascularization and regeneration. Nat Med. 2003 Jun;9(6):702-12. doi: 10.1038/nm0603-702. PMID 12778169
- [Background] Falanga V, Iwamoto S, Chartier M, Yufit T, Butmarc J, Kouttab N, Shrayer D, Carson P. Autologous bone marrow-derived cultured mesenchymal stem cells delivered in a fibrin spray accelerate healing in murine and human cutaneous wounds. Tissue Eng. 2007 Jun;13(6):1299-312. doi: 10.1089/ten.2006.0278. PMID 17518741
- [Background] Kirana S, Stratmann B, Lammers D, Negrean M, Stirban A, Minartz P, Koerperich H, Gastens MH, Gotting C, Prohaska W, Kleesiek K, Tschoepe D. Wound therapy with autologous bone marrow stem cells in diabetic patients with ischaemia-induced tissue ulcers affecting the lower limbs. Int J Clin Pract. 2007 Apr;61(4):690-2. doi: 10.1111/j.1742-1241.2007.01303.x. PMID 17394441
- [Background] Dash NR, Dash SN, Routray P, Mohapatra S, Mohapatra PC. Targeting nonhealing ulcers of lower extremity in human through autologous bone marrow-derived mesenchymal stem cells. Rejuvenation Res. 2009 Oct;12(5):359-66. doi: 10.1089/rej.2009.0872. PMID 19929258
- [Background] Horwitz EM, Gordon PL, Koo WK, Marx JC, Neel MD, McNall RY, Muul L, Hofmann T. Isolated allogeneic bone marrow-derived mesenchymal cells engraft and stimulate growth in children with osteogenesis imperfecta: Implications for cell therapy of bone. Proc Natl Acad Sci U S A. 2002 Jun 25;99(13):8932-7. doi: 10.1073/pnas.132252399. PMID 12084934
- [Background] Strauer BE, Brehm M, Zeus T, Kostering M, Hernandez A, Sorg RV, Kogler G, Wernet P. Repair of infarcted myocardium by autologous intracoronary mononuclear bone marrow cell transplantation in humans. Circulation. 2002 Oct 8;106(15):1913-8. doi: 10.1161/01.cir.0000034046.87607.1c. PMID 12370212
- [Background] Chen SL, Fang WW, Ye F, Liu YH, Qian J, Shan SJ, Zhang JJ, Chunhua RZ, Liao LM, Lin S, Sun JP. Effect on left ventricular function of intracoronary transplantation of autologous bone marrow mesenchymal stem cell in patients with acute myocardial infarction. Am J Cardiol. 2004 Jul 1;94(1):92-5. doi: 10.1016/j.amjcard.2004.03.034. PMID 15219514
- [Background] Lunde K, Solheim S, Aakhus S, Arnesen H, Abdelnoor M, Egeland T, Endresen K, Ilebekk A, Mangschau A, Fjeld JG, Smith HJ, Taraldsrud E, Grogaard HK, Bjornerheim R, Brekke M, Muller C, Hopp E, Ragnarsson A, Brinchmann JE, Forfang K. Intracoronary injection of mononuclear bone marrow cells in acute myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1199-209. doi: 10.1056/NEJMoa055706. PMID 16990383
- [Background] Fuchs S, Kornowski R, Weisz G, Satler LF, Smits PC, Okubagzi P, Baffour R, Aggarwal A, Weissman NJ, Cerqueira M, Waksman R, Serrruys P, Battler A, Moses JW, Leon MB, Epstein SE. Safety and feasibility of transendocardial autologous bone marrow cell transplantation in patients with advanced heart disease. Am J Cardiol. 2006 Mar 15;97(6):823-9. doi: 10.1016/j.amjcard.2005.09.132. Epub 2006 Jan 30. PMID 16516583
- [Background] Rubio D, Garcia-Castro J, Martin MC, de la Fuente R, Cigudosa JC, Lloyd AC, Bernad A. Spontaneous human adult stem cell transformation. Cancer Res. 2005 Apr 15;65(8):3035-9. doi: 10.1158/0008-5472.CAN-04-4194. PMID 15833829 (Retraction: PMID 20710046 de la Fuente R, Bernad A, Garcia-Castro J, Martin MC, Cigudosa JC. Cancer Res. 2010 Aug 15;70(16):6682)
- [Background] Bernardo ME, Zaffaroni N, Novara F, Cometa AM, Avanzini MA, Moretta A, Montagna D, Maccario R, Villa R, Daidone MG, Zuffardi O, Locatelli F. Human bone marrow derived mesenchymal stem cells do not undergo transformation after long-term in vitro culture and do not exhibit telomere maintenance mechanisms. Cancer Res. 2007 Oct 1;67(19):9142-9. doi: 10.1158/0008-5472.CAN-06-4690. PMID 17909019
- [Background] Miura Y, Gao Z, Miura M, Seo BM, Sonoyama W, Chen W, Gronthos S, Zhang L, Shi S. Mesenchymal stem cell-organized bone marrow elements: an alternative hematopoietic progenitor resource. Stem Cells. 2006 Nov;24(11):2428-36. doi: 10.1634/stemcells.2006-0089. PMID 17071859
- [Background] Dahl JA, Duggal S, Coulston N, Millar D, Melki J, Shahdadfar A, Brinchmann JE, Collas P. Genetic and epigenetic instability of human bone marrow mesenchymal stem cells expanded in autologous serum or fetal bovine serum. Int J Dev Biol. 2008;52(8):1033-42. doi: 10.1387/ijdb.082663jd. PMID 18956336
- [Background] Tarte K, Gaillard J, Lataillade JJ, Fouillard L, Becker M, Mossafa H, Tchirkov A, Rouard H, Henry C, Splingard M, Dulong J, Monnier D, Gourmelon P, Gorin NC, Sensebe L; Societe Francaise de Greffe de Moelle et Therapie Cellulaire. Clinical-grade production of human mesenchymal stromal cells: occurrence of aneuploidy without transformation. Blood. 2010 Feb 25;115(8):1549-53. doi: 10.1182/blood-2009-05-219907. Epub 2009 Dec 23. PMID 20032501
- [Background] Rosland GV, Svendsen A, Torsvik A, Sobala E, McCormack E, Immervoll H, Mysliwietz J, Tonn JC, Goldbrunner R, Lonning PE, Bjerkvig R, Schichor C. Long-term cultures of bone marrow-derived human mesenchymal stem cells frequently undergo spontaneous malignant transformation. Cancer Res. 2009 Jul 1;69(13):5331-9. doi: 10.1158/0008-5472.CAN-08-4630. Epub 2009 Jun 9. PMID 19509230
- [Background] Garcia S, Bernad A, Martin MC, Cigudosa JC, Garcia-Castro J, de la Fuente R. Pitfalls in spontaneous in vitro transformation of human mesenchymal stem cells. Exp Cell Res. 2010 May 15;316(9):1648-50. doi: 10.1016/j.yexcr.2010.02.016. Epub 2010 Feb 18. No abstract available. PMID 20171963
- [Background] Prockop DJ, Brenner M, Fibbe WE, Horwitz E, Le Blanc K, Phinney DG, Simmons PJ, Sensebe L, Keating A. Defining the risks of mesenchymal stromal cell therapy. Cytotherapy. 2010 Sep;12(5):576-8. doi: 10.3109/14653249.2010.507330. PMID 20735162
- [Background] Ladwig GP, Robson MC, Liu R, Kuhn MA, Muir DF, Schultz GS. Ratios of activated matrix metalloproteinase-9 to tissue inhibitor of matrix metalloproteinase-1 in wound fluids are inversely correlated with healing of pressure ulcers. Wound Repair Regen. 2002 Jan-Feb;10(1):26-37. doi: 10.1046/j.1524-475x.2002.10903.x. PMID 11983004
- [Background] Mast BA, Schultz GS. Interactions of cytokines, growth factors, and proteases in acute and chronic wounds. Wound Repair Regen. 1996 Oct;4(4):411-20. doi: 10.1046/j.1524-475X.1996.40404.x. PMID 17309691